CLINICAL TRIAL: NCT05207878
Title: Interhemispheric Communication and Compensation in Peripheral Nerve Injury
Brief Title: Interhemispheric Connectivity and Compensation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 202009183; R01NS114046-01A1 (NIH)
Record Dates: First submitted 2021-12-25; First posted 2022-01-26 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Peripheral Nerve Injury Upper Limb; Healthy
Keywords: laterality of motor control; movement; functional magnetic resonance imaging; functional laterality

STUDY DESIGN:
Intervention Model Description: The only "intervention" is the movement task. All participants receive the same task.
Masking Description: During TMS, participants will be masked to whether they receive effective or sham stimulation on a given trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Movement task (Experimental): All participants perform the STEGA-MRI (standardized tracing evaluation & grapheme assessment - MRI) precision drawing task during fMRI scanning.
  Motor assessments outside the MRI do not qualify as interventions.
  Interventions: Other: STEGA-MRI

INTERVENTIONS:
Other: STEGA-MRI — Precision drawing task (movement assessment)

SUMMARY:
The goal of this study is to determine which parts of the brain make it possible for some people to move skillfully with their left non-dominant hand.

DETAILED DESCRIPTION:
This is a one-visit study, in which right-handed participants (individuals with unilateral peripheral nerve injury to the right upper limb, and healthy controls) will complete surveys and perform movement tasks. Movement tasks will be performed inside and outside a magnetic resonance imaging (MRI) scanner.

Some participants will also receive transcranial magnetic stimulation (TMS) to briefly interfere with these putative brain networks.

ELIGIBILITY:
This study contains two groups: typical controls and patients. Participants will be matched by age and sex between the two groups. No randomization will occur.

A. Inclusion criteria (all participants):

1. Age ≥ 18
2. English speaking and reading
3. Able to fit in Prisma scanner bore (60 cm diameter)
4. Right hand dominant (self report, and Edinburgh handedness ≥ +40)

B. Inclusion criteria (patients only):

1. Chronic unilateral upper extremity peripheral nerve injury to the right side

   * "Chronic" defined as ≥ 6 months since injury
   * "Upper extremity" defined as hand, arm, or shoulder (including e.g. brachial plexus)
   * "Injury" defined as localized cause (e.g. mechanical/tumor, not distributed pathology), including compression
2. Some impairment to writing, requiring both of:

   * Difficulty writing, as determined by score 2+ (Mild+) on "How much difficulty have you had in the last week with writing?" (From Disabilities of the Arm, Shoulder, and Hand survey question #2)
   * Box and Blocks motor performance ≥1 standard deviation below the mean of age-matched healthy adults (Mathiowetz et al. 1985, AJOT).

C. Exclusion criteria (all participants)

1. Currently intoxicated or otherwise non-compliant
2. Chronic pain diagnosis unrelated to the nerve injury
3. Uncorrected visual impairment that interferes with ability to see drawings in MRI
4. Motor function diagnoses that affect function of the left hand, now or in past 2 years
5. Motor function diagnoses currently affecting the right hand, unrelated to the nerve injury

   * This is not meant to exclude a single event with complex consequences (e.g. nerve and tendon)
   * This is not meant to exclude multiple nerve injuries in the same arm, if each one is eligible (II.B.1)
   * This is meant to exclude e.g. injury and unrelated musculoskeletal disorder in same arm
6. Upper extremity surgery, including peripheral nerve surgery, within last 2 months
7. Contraindication for MRI
8. Contraindication for transcranial magnetic stimulation (TMS)

   * May exclude from TMS only (since not all participants undergo TMS), or exclude from full study
9. Amputation affecting any part of thumb, index, or middle fingers (including higher level, e.g. whole hand)
10. History of chronic cocaine use (based on medical record or volunteered; will not actively inquire)
11. Diagnosis of schizophrenia or other rare psychiatric disorder

    * This is not meant to exclude depression or anxiety
12. History of major neurological diagnosis, e.g. stroke, traumatic brain injury, Alzheimer's, Parkinson's

    * This is not meant to exclude concussion UNLESS < 6 months ago, or post-concussion syndrome (diagnosed or self-report)

D. Exclusion criteria (controls only)

1. Motor function diagnoses that affect function of either hand, now or in past 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
BOLD (blood oxygen level dependent) signal in ROIs (regions of interest) | Day 1
  BOLD signal in key ROIs (primary motor and posterior parietal cortex). ROI selection may be revisited after preliminary data review (35 participants)

SECONDARY OUTCOMES:
Drawing smoothness | Day 1
  Velocity smoothness in STEGA-MRI (Standardized Tracing Evaluation and Grapheme Assessment - MRI version) task
Hand choice | Day 1
  Percentage of grasps made with right hand

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin A Philip, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
For participants who consent to us sharing their data with other researchers, we will share all anonymized data (behavioral, survey, and MRI), including data dictionaries.
  Note that this clinical trial is a "prospective basic science study involving human participants;" i.e., a study that falls within the NIH definition of clinical trial while also meeting the definition of basic research.
Supporting Information: Study Protocol, ICF
Time Frame: Will become available after summary data are published. Will remain available indefinitely.

DOCUMENTS (1):
  • Informed Consent Form (2024-03-20): https://cdn.clinicaltrials.gov/large-docs/78/NCT05207878/ICF_001.pdf